CLINICAL TRIAL: NCT07179237
Title: Evaluation of the Efficacy of Carminal on the Gastric Mucosa in Patients With Helicobacter Pylori Positive Gastritis
Brief Title: Efficacy of Carminal in Helicobacter Pylori Gastritis
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Catalysis SL (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: CARMINAL_HPYLORI_SERBIA2025
Record Dates: First submitted 2025-09-09; First posted 2025-09-17 (Actual); Last update posted 2025-09-17 (Actual); Status verified 2025-09

CONDITIONS: H Pylori Gastritis; H Pylori Infection; H Pylori Eradication; Gastritis Associated With Helicobacter Pylori; Gastric Mucosal Lesion
Keywords: Antioxidant; Aloe vera; Food Supplement; Helicobacter Pylori; Gastritis; Gastric mucosa
MeSH Terms: conditions — Gastritis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Carminal Group (Experimental): Participants in this arm (n=40) will receive:
  Carminal oral solution, 30 ml once daily (1 vial BID), administered for 14 days during standard Helicobacter pylori eradication therapy.
  Following successful eradication, Carminal treatment will continue for 12 additional weeks.
  Carminal is a supplement containing Aloe vera extract, olive extract, glutamic acid, zinc, and other components with potential antioxidant, anti-inflammatory, and immunomodulatory effects on gastric mucosa.
  The intervention aims to support mucosal recovery post-eradication and improve dyspeptic symptoms.
  Interventions: Dietary Supplement: Carminal Oral solution
- Placebo Group (Placebo Comparator): Participants in this arm (n=40) will receive:
  Placebo, matched in appearance and administration schedule to Carminal, for 14 days during standard H. pylori eradication therapy.
  Following successful eradication, placebo treatment will continue for 12 additional weeks.
  This arm serves as the control group to evaluate the efficacy of Carminal in mucosal recovery and symptom improvement.
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: Carminal Oral solution — Carminal is an oral dietary supplement presented in 30 ml vials, administered once daily (1 vial BID). It contains Aloe vera extract, olive extract, glutamic acid, zinc, and other components with potential antioxidant, anti-inflammatory, and immunomodulatory effects on gastric mucosa. In this study, Carminal is administered for 14 days during standard Helicobacter pylori eradication therapy, followed by 12 weeks of continued treatment post-eradication to support mucosal recovery and improve dyspeptic symptoms.
  Other Names: Carminal; Carminal supplement; Carminal 30 ml vials
  Arms: Carminal Group
Other: Placebo — Placebo is an oral solution presented in 30 ml vials, identical in appearance, taste, color, and smell to Carminal, but without any active ingredients. It is administered once daily (1 vial BID) for 14 days during standard Helicobacter pylori eradication therapy, followed by 12 weeks of continued placebo treatment post-eradication. This comparator is used to evaluate the efficacy of Carminal in mucosal recovery and symptom improvement in patients with H. pylori positive gastritis.
  Other Names: Carminal Placebo; Placebo 30 ml vials
  Arms: Placebo Group

SUMMARY:
Eighty patients will be included and randomized in two groups, one group (40 patients) will be administered 30 ml of the supplement Carminal, once a day, plus therapy for HP gastitis and the control group (40 patients) will be given standard therapy for HP gastritis with placebo. Treatment will begin after complection of upper endoscopy with histology results from biopted gastric mucosa. Treatment with Carminal will be continued after successful HP eradication during 12 weeks. The final evaluation will take place 12 weeks after the last Carminal intake, when control endoscopy with histology will be performed. The study will last approximately 24 weeks.

DETAILED DESCRIPTION:
Helicobacter pylori-induced gastritis is an infectious disease based on objective pathological criteria. After the successful eradication of the infection, the recovery of the mucosa occurs through a gradual process that lasts several months. HP eradication is a therapeutic modality for the treatment of non-atrophic gastritis, and it leads to the regression of atrophic gastritis and the reduction of the risk of gastric cancer. In patients with histologically verified intestinal metaplasia, HP eradication does not reduce the risk of malignancy, but reduces inflammation and atrophy, thereby slowing its further progression. It is considered that advanced changes of the mucosa are not fully reversible, while even atrophy can be reversible in certain cases. There are controversial data about reversibility of intestinal metaplasia. However, HP treatment is challenged by the continuously rising antibiotic resistance and demands for susceptibility testing with consideration of novel molecular technologies and careful selection of first line and rescue therapies. On the other hand, the role of HP and antibiotic therapies and their impact on the gut microbiota are also considered.

The Aloe vera plant (Aloe vera) is a well-known natural substance with several advantages. Aloe vera is frequently utilized as a fundamental component in medications and cosmetics, either directly or after being processed with additional substances. Aloe vera is a member of the Liliaceae family, which has over 200 species. Multiple preclinical studies have demonstrated that ingesting aloe vera juice in specific amounts may contribute to healing stomach ulcers and may be a natural cure for heartburn. Additionally, according to experimental studies aloe vera has the capacity to increase the production of pepsin, a stomach enzyme that aids in digestion. These findings suggest that using a combination of aloe vera with additional substances can have a synergistic antinflammatory and immunomodulatory effect in vivo on gastric mucosa and peptic ulcer disease on animal models.

Carminal, produced by Laboratorios Catalysis, S. L., is an oral solution and supplement that combines aloe vera extract and various substances known for their potential antioxidant, anti-inflammatory and immunomodulatory properties on gastric mucosa.

The goal of this study is to assess how Carminal affects the HP eradication and recovery of gastric mucosa after successful HP eradication and effect on related symptoms.

The trial will be conducted in accordance with the protocol, Good Clinical Practice (GCP) and in compliance with the regulations in force in the Republic of Serbia.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18 years or older
* Patients with clinical symptoms of dyspepsia
* Patients diagnosed with Helicobacter pylori positive gastritis, confirmed by upper endoscopy with histology
* Patients who give written informed consent to participate in the study

Exclusion Criteria:

* Patients with peptic ulcer disease
* Patients with previous gastric surgery
* Patients with current malignancy or the history of any previous malignancies
* Patients taking another investigational product, or have taken any investigational product in the last year
* Patients with known hypersensitivity to any ingredients found in the investigational product.
* Decompensated intercurrent illnesses, including: active infections, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, liver disease, and psychiatric illnesses that may limit adherence to the requirements of the clinical trial, or any other special condition that, according to the physician's judgement, jeopardises the patient's health or life during participation in the trial.
* Planned pregnancy for the duration of trial, pregnancy, breast feeding, or postpartum period.
* Patients with human immunodeficiency virus (HIV).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2025-08-04 (Actual); Primary Completion 2026-08-03 (Estimated); Study Completion 2026-10-05 (Estimated)

PRIMARY OUTCOMES:
Glasgow Dyspepsia Severity Score | Baseline, Week 7 (post-eradication), Week 20 (end of treatment)
  Change in dyspeptic symptoms assessed using the Glasgow Dyspepsia Severity Score questionnaire at baseline, after eradication therapy, and at the end of Carminal/placebo treatment.
Endoscopic assessment of gastric mucosa | Baseline and Week 21
  Endoscopic evaluation of gastric mucosa performed before treatment and at the end of the study to assess mucosal recovery, including presence of gastritis, intestinal metaplasia, and other morphological changes.
Histological assessment of gastric mucosa | Baseline and Week 21
  Histological analysis of gastric biopsies to evaluate inflammation, atrophy, foveolar hyperplasia, and intestinal metaplasia before and after treatment.

SECONDARY OUTCOMES:
Leeds Dyspepsia Score | Baseline, Week 7, Week 20
  Change in dyspeptic symptoms assessed using the Leeds Dyspepsia Score questionnaire at baseline, after eradication therapy, and at the end of treatment.
Helicobacter pylori status (HP antigen stool test) | Week 7
  HP antigen presence in stool samples to confirm eradication success after 14-day standard therapy.
Patient satisfaction after treatment completion | Week 20
  Patient-reported satisfaction with treatment outcomes collected via questionnaire at the end of the study.
Occurrence of adverse events | Throughout the study (Week 1 to Week 21)
  Monitoring and recording of any adverse events (AEs), including type, duration, intensity, seriousness, and outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Dragana Mijač, MD, PhD, Principal Investigator — Clinic for Gastroenterohepatology, Clinical Center of Serbia
Locations (2):
- Serbia (2):
  - Clinical Center of Serbia - Clinic for Gastroenterohepatology, Belgrade, Central Serbia
  - Zvezdara Medical Center - Department of Gastroenterology, Belgrade, Central Serbia

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: CSR

REFERENCES:
- [Background] Dixon MF, Genta RM, Yardley JH, Correa P. Classification and grading of gastritis. The updated Sydney System. International Workshop on the Histopathology of Gastritis, Houston 1994. Am J Surg Pathol. 1996 Oct;20(10):1161-81. doi: 10.1097/00000478-199610000-00001. PMID 8827022
- [Background] Sugano K, Tack J, Kuipers EJ, Graham DY, El-Omar EM, Miura S, Haruma K, Asaka M, Uemura N, Malfertheiner P; faculty members of Kyoto Global Consensus Conference. Kyoto global consensus report on Helicobacter pylori gastritis. Gut. 2015 Sep;64(9):1353-67. doi: 10.1136/gutjnl-2015-309252. Epub 2015 Jul 17. PMID 26187502
- [Background] Malfertheiner P, Megraud F, Rokkas T, Gisbert JP, Liou JM, Schulz C, Gasbarrini A, Hunt RH, Leja M, O'Morain C, Rugge M, Suerbaum S, Tilg H, Sugano K, El-Omar EM; European Helicobacter and Microbiota Study group. Management of Helicobacter pylori infection: the Maastricht VI/Florence consensus report. Gut. 2022 Aug 8:gutjnl-2022-327745. doi: 10.1136/gutjnl-2022-327745. Online ahead of print. PMID 35944925
- [Background] Wang C, Yuan Y, Hunt RH. The association between Helicobacter pylori infection and early gastric cancer: a meta-analysis. Am J Gastroenterol. 2007 Aug;102(8):1789-98. doi: 10.1111/j.1572-0241.2007.01335.x. Epub 2007 May 23. PMID 17521398
- [Background] Graham DY. History of Helicobacter pylori, duodenal ulcer, gastric ulcer and gastric cancer. World J Gastroenterol. 2014 May 14;20(18):5191-204. doi: 10.3748/wjg.v20.i18.5191. PMID 24833849
- [Background] Liou JM, Fang YJ, Chen CC, Bair MJ, Chang CY, Lee YC, Chen MJ, Chen CC, Tseng CH, Hsu YC, Lee JY, Yang TH, Luo JC, Chang CC, Chen CY, Chen PY, Shun CT, Hsu WF, Hu WH, Chen YN, Sheu BS, Lin JT, Wu JY, El-Omar EM, Wu MS; Taiwan Gastrointestinal Disease and Helicobacter Consortium. Concomitant, bismuth quadruple, and 14-day triple therapy in the first-line treatment of Helicobacter pylori: a multicentre, open-label, randomised trial. Lancet. 2016 Nov 12;388(10058):2355-2365. doi: 10.1016/S0140-6736(16)31409-X. Epub 2016 Oct 18. PMID 27769562
- [Background] Hooi JKY, Lai WY, Ng WK, Suen MMY, Underwood FE, Tanyingoh D, Malfertheiner P, Graham DY, Wong VWS, Wu JCY, Chan FKL, Sung JJY, Kaplan GG, Ng SC. Global Prevalence of Helicobacter pylori Infection: Systematic Review and Meta-Analysis. Gastroenterology. 2017 Aug;153(2):420-429. doi: 10.1053/j.gastro.2017.04.022. Epub 2017 Apr 27. PMID 28456631